CLINICAL TRIAL: NCT07300306
Title: Validation of the SOFA-2 Score for 30-Day Mortality in Intensive Care Units in Turkey and Determination of Sepsis-3 Prevalence - A Multicenter Hybrid Observational Study.
Brief Title: Validation of SOFA-2 for Mortality and Sepsis-3 Prevalence in Turkey
Acronym: TURK-SOFA2
Status: Not yet recruiting | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Mustafa Kemal Arslantas, Professor of Anesthesiology and Anesthesiology and Reanimation, Marmara University
Other Study IDs: TURK-SOFA2; 09.2025.25-1065 (Other: Marmara University School of Medicine)
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Sepsis; Septic Shock; Critical Illness; Organ Dysfunction
Keywords: SOFA-2 Score; Sepsis-3; Intensive Care Unit; Mortality Prediction; Organ Failure Assessment; Validation Study
MeSH Terms: conditions — Sepsis; Shock, Septic; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary Validation Cohort: Adult patients admitted to the ICU during the 7-day prospective recruitment window. Organ dysfunction scores are calculated within the first 24 hours to validate SOFA-2 for 30-day mortality.
- Point Prevalence Cohort: All adult patients present in the ICU on the designated single "Index Day" (08:00 to 08:00). Used specifically to determine the point prevalence of Sepsis-3 and septic shock.

SUMMARY:
The goal of this observational study is to validate the effectiveness of the new SOFA-2 score in predicting mortality and to determine the current frequency of sepsis in adult patients admitted to Intensive Care Units (ICUs) in Turkey. The main questions it aims to answer are:

* Does the SOFA-2 score accurately predict 30-day mortality in ICU patients?
* What is the prevalence of Sepsis-3 and septic shock in Turkish ICUs?

Researchers will compare the new SOFA-2 score to the existing SOFA-1 score to see if the new score provides better predictive accuracy for patient outcomes.

Participants will not receive any experimental intervention. Researchers will collect data from routine medical care, including:

* Vital signs, laboratory test results, and details of organ support (such as mechanical ventilation or dialysis) during the first 24 hours of admission.
* Survival status at 30 days.

DETAILED DESCRIPTION:
Background and Rationale Sepsis remains a leading cause of mortality in Intensive Care Units (ICUs) globally. The operational definition of sepsis (Sepsis-3) relies on the Sequential Organ Failure Assessment (SOFA) score. However, the original SOFA score, developed in 1996, predates modern critical care interventions such as High-Flow Nasal Cannula (HFNC), non-invasive ventilation, and contemporary vasopressor strategies. Consequently, the original score has limitations in accurately characterizing organ dysfunction in the modern ICU setting.

The recently updated SOFA-2 score (JAMA, 2025) addresses these shortcomings by revising scoring thresholds and incorporating modern respiratory and cardiovascular support modalities. While validated in large international cohorts, the SOFA-2 score requires local validation in Turkey to account for regional differences in patient demographics, genetics, and healthcare infrastructure before widespread clinical adoption.

Study Design This is a multicenter, prospective, hybrid observational study comprising two distinct components to maximize data utility while minimizing data collection burden:

Prospective Validation Cohort (Primary): A 7-day recruitment window will be established (e.g., January 2026). During this period, all consecutive adult patients (aged 18 and older) admitted to participating ICUs will be enrolled. Baseline organ dysfunction scores will be calculated using the worst physiological values recorded during the first 24 hours of admission. These patients will be followed up for 30-day all-cause mortality to validate the predictive performance (discrimination and calibration) of the SOFA-2 score compared to the original SOFA-1 score.

Point-Prevalence Cohort (Secondary): Within the 7-day window, a specific 24-hour period will be designated as the "Index Day." This cross-sectional component will include all patients present in the ICU at 08:00 AM on the index day, plus any new admissions over the subsequent 24 hours. This cohort will be used specifically to determine the point prevalence of Sepsis-3 and septic shock in Turkish ICUs, providing a snapshot of the current epidemiological burden compared to historical data.

Data Collection Methodology To ensure standardization and eliminate inter-rater variability, participating centers will not manually calculate scores. Instead, researchers will record raw physiological, laboratory, and therapeutic variables (e.g., PaO2, platelet count, exact vasopressor doses, Glasgow Coma Scale) into a central electronic Case Report Form (eCRF). The study algorithms will then centrally and automatically calculate SOFA-1, SOFA-2, APACHE II, and Sepsis-3 status for all patients. This approach ensures that the comparison between scoring systems is objective and mathematically consistent.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older.
* Admitted to the Intensive Care Unit (ICU) during the specified study recruitment window.
* For the Validation Cohort: Patients staying in the ICU for at least 24 hours.
* For the Point Prevalence Cohort: Patients present in the ICU at 08:00 AM on the designated "Index Day" or admitted within the subsequent 24 hours.

Exclusion Criteria:

* Patients younger than 18 years of age.
* Patients admitted to Pediatric Intensive Care Units.
* Patients admitted to Coronary Care Units (CCU).
* Patients admitted to Cardiovascular Surgery Intensive Care Units.
* Patients admitted solely for the purpose of organ donation.
* Patients with missing core data components required for score calculation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (aged 18 years or older) admitted to adult Intensive Care Units (ICUs) in participating University Hospitals, Training and Research Hospitals, State Hospitals, and Private Hospitals across Turkey. The population includes consecutive admissions with various critical illness etiologies, excluding those admitted to coronary or cardiovascular surgery units.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
0-Day All-Cause Mortality | 30 days
  The vital status (alive or dead) of patients assessed at 30 days post-ICU admission. This measure is used to validate the predictive accuracy (discrimination and calibration) of the SOFA-2 score.

SECONDARY OUTCOMES:
Point Prevalence of Sepsis-3 | Index Day (24 hours)
  The proportion of patients meeting the Third International Consensus Definitions for Sepsis (Sepsis-3) in the ICU on the designated index day.

OTHER OUTCOMES:
Vasopressor-Free Days (VFD-28) | 28 days
  The number of days alive and free of vasopressor therapy within the first 28 days following admission.
Length of ICU Stay | From date of admission until the date of discharge or death, assessed up to 90 days.
  The duration of stay in the Intensive Care Unit from admission to discharge or death.
Length of Hospital Stay | From date of admission until the date of discharge or death, assessed up to 90 days.
  The total duration of hospitalization from admission to discharge or death.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University Pendik Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ranzani OT, Singer M, Salluh JIF, Shankar-Hari M, Pilcher D, Berger-Estilita J, Coopersmith CM, Juffermans NP, Laffey J, Reinikainen M, Neto AS, Tavares M, Timsit JF, Arias Lopez MDP, Arulkumaran N, Aryal D, Azoulay E, Celi LA, Chaudhuri D, De Lange D, De Waele J, Dos Santos CC, Du B, Einav S, Engelbrecht T, Fazla F, Ferrer R, Finazzi S, Fujii T, Gershengorn HB, Greene JD, Haniffa R, Hao S, Hasan MS, Hollenberg S, Ippolito M, Jung C, Kirov M, Kobari S, Lakbar I, Lipman J, Liu V, Liu X, Lobo SM, Magatti D, Martin GS, Metnitz B, Metnitz P, Myatra SN, Oczkowski S, Paiva JA, Paruk F, Pekkarinen PT, Piquilloud L, Polkki A, Prescott HC, Blaser AR, Rezende E, Robba C, Rochwerg B, Ruckly S, Samei R, Schenck EJ, Secombe P, Sendagire C, Siaw-Frimpong M, Simpkin AJ, Soares M, Summers C, Szczeklik W, Takala J, Tanaka S, Tricella G, Vincent JL, Wendon J, Zampieri FG, Rhodes A, Moreno R. Development and Validation of the Sequential Organ Failure Assessment (SOFA)-2 Score. JAMA. 2025 Dec 16;334(23):2090-2103. doi: 10.1001/jama.2025.20516. PMID 41159833
- [Result] Weijs PJM. Route, early or energy? ... Protein improves protein balance in critically ill patients. Crit Care. 2018 Apr 14;22(1):91. doi: 10.1186/s13054-018-2015-z. No abstract available. PMID 29653538
- See also: Related Info — https://sepsis.tr/